CLINICAL TRIAL: NCT01945866
Title: Short-term Evaluation of Combination Corticosteroid+Anti-VEGF Treatment for Persistent Central-Involved Diabetic Macular Edema Following Anti-VEGF Therapy
Brief Title: Phase II Combination Steroid and Anti-VEGF for Persistent DME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Allergan (Industry); Genentech, Inc. (Industry); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRCR.net Protocol U; EY14231 (Other Grant/Funding Number: National Eye Institute); EY23207 (Other Grant/Funding Number: National Eye Institute); EY18817 (Other Grant/Funding Number: National Eye Institute)
Record Dates: First submitted 2013-09-12; First posted 2013-09-19 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Anti-vascular endothelial growth factor; Dexamethasone Intravitreal implant; Ranibizumab intravitreal injection
MeSH Terms: interventions — Ranibizumab; Dexamethasone; Calcium Dobesilate; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham + intravitreal ranibizumab 0.3 mg (Active Comparator): Intravitreal ranibizumab will be given on the day of randomization. The sham injection will be given within 0-8 days of the ranibizumab injection. If the injections are given consecutively on the same day, the sham injection must be given first. Follow-up intravitreal injections of ranibizumab will be given up to every 4 weeks using defined treatment criteria.
  Interventions: Drug: intravitreal ranibizumab 0.3 mg; Procedure: Sham injection
- Intravitreal dexamethasone+intravitreal ranibizumab 0.3mg (Experimental): The initial intravitreal ranibizumab injection will be given on the day of randomization. The dexamethasone intravitreal injection will be given within 0-8 days of the ranibizumab injection. If defined criteria are met, a second dexamethasone injection in combination with intravitreal ranibizumab (within 0-8 days) will be given at the 12 week visit. If the injections are given consecutively on the same day, the ranibizumab injection must be given first.
  Interventions: Drug: intravitreal ranibizumab 0.3 mg; Drug: dexamethasone intravitreal implant

INTERVENTIONS:
Drug: intravitreal ranibizumab 0.3 mg — Intravitreal injection of 0.3mg ranibizumab performed on the day of randomization and up to every 4 weeks using defined treatment criteria
  Other Names: Lucentis
Drug: dexamethasone intravitreal implant — The dexamethasone intravitreal injection will be given within 0-8 days of the ranibizumab injection. If defined criteria are met, a second dexamethasone injection in combination with intravitreal ranibizumab (within 0-8 days) will be given at the 12 week visit. If the injections are given consecutively on the same day, the ranibizumab injection must be given first.
  Other Names: Ozurdex
  Arms: Intravitreal dexamethasone+intravitreal ranibizumab 0.3mg
Procedure: Sham injection — No injection is given. It is a sham injection to keep the participant masked. The sham injection will be given within 0-8 days of the ranibizumab injection. If the injections are given consecutively on the same day, the sham injection must be given first.
  Arms: Sham + intravitreal ranibizumab 0.3 mg

SUMMARY:
Although anti-vascular endothelial growth factor (VEGF) therapy is generally effective as treatment for center-involved diabetic macular edema (DME), a substantial proportion of anti-VEGF-treated eyes with DME do not achieve vision of 20/20 or complete resolution of retinal thickening. Indeed, over 50% of ranibizumab-treated eyes did not achieve a 2 or more line improvement in visual acuity from baseline at 2 years in Protocol I, a previous DRCR.net (Diabetic Retinopathy Clinical Research Network) study. Furthermore, 27% of ranibizumab-treated eyes still had central subfield (CSF) thickness on time-domain optical coherence tomography (OCT) ≥ 300 at 1 year, and more than 40% of ranibizumab-treated eyes did not achieve complete resolution of retinal thickening (< 250 microns) by 2 years. Thus, there is a need for alternative or additional treatments that will improve vision by reducing retinal edema in eyes with persistent DME following previous anti-VEGF therapy. Intravitreal steroid is not as efficacious as ranibizumab in eyes with DME overall, but it has been shown to have a positive effect for DME in some eyes and might add benefit in eyes that are already receiving anti-VEGF.

The main objective of this study is to assess the short-term effects of combination steroid+anti-VEGF therapy on visual acuity and retinal thickness on OCT in comparison with that of continued anti-VEGF therapy alone in eyes with persistent central-involved DME and visual acuity impairment despite previous anti-VEGF treatment. This study will provide important information for the design of a future confirmatory phase III clinical trial on the efficacy of combination steroid and anti-VEGF in eyes with persistent DME and vision impairment following previous anti-VEGF therapy. The primary outcome for efficacy will be the mean change in visual acuity at 24 weeks.

Each study eye is required to complete a 12-week run-in phase. The run-in phase will identify study eyes that truly have persistent DME despite anti-VEGF therapy by requiring an additional 3 injections while also collecting standardized visual acuity and OCT measurements. At the enrollment, 4-week and 8-week visits of the run-in phase, enrolled eyes will receive an intravitreal injection of ranibizumab 3mg. Then at the 12-week run-in visit, if the eye still has persistent DME, it will be randomized to receive either intravitreal sham+intravitreal ranibizumab 0.3 or intravitreal dexamethasone+intravitreal ranibizumab 0.3 injections. The randomized study duration is 24 week, during which a protocol visit takes place every month. The combination injections of sham+ranibizumab or dexamethasone +ranibizumab will be given at the randomization visit (baseline) and at the 12-week visit after randomization. In between, an intravitreal injection of ranibizumab only will be given to study eyes at the 4, 8, 16 and 20 week visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years i) Individuals <18 years old are not being included because DME is so rare in this age group that the diagnosis of DME may be questionable.
2. Diagnosis of diabetes mellitus (type 1 or type 2)
3. Any one of the following will be considered to be sufficient evidence that diabetes is present:

   1. Current regular use of insulin for the treatment of diabetes
   2. Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
   3. Documented diabetes by ADA (American Diabetes Association) and/or WHO (World Health Organization) criteria
4. At least one eye meets the study eye criteria listed below.
5. Fellow eye (if not a study eye) meets criteria.
6. Able and willing to provide informed consent.

Meets all of the following ocular criteria in at least the one eye:

1. At least 3 injections of anti-VEGF drug (ranibizumab, bevacizumab, or aflibercept) within the prior 20 weeks.
2. Visual acuity letter score in study eye ≤ 78 and ≥24 (approximate Snellen equivalent 20/32 to 20/320).
3. On clinical exam, definite retinal thickening due to DME involving the center of the macula.
4. OCT CSF thickness, within 8 days of enrollment:

   i) On Zeiss Cirrus ≥ 290 microns in women; ≥ 305 in men ii) On Heidelberg Spectralis: ≥ 305 microns in women; ≥ 320 in men
5. Media clarity, pupillary dilation, and individual cooperation sufficient for adequate OCTs.

Exclusion Criteria:

An individual is not eligible if any of the following exclusion criteria are present:

1. History of chronic renal failure requiring dialysis or kidney transplant.
2. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
3. Initiation of intensive insulin treatment (a pump or multiple daily injections) within 4 months prior to randomization or plans to do so in the next 4 months.
4. Participation in an investigational trial within 30 days of enrollment that involved treatment with any drug that has not received regulatory approval for the indication being studied. Note: study participants cannot receive another investigational drug while participating in the study.
5. Known allergy to any component of the study drugs (including povidone iodine prep).
6. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, the individual can become eligible.
7. Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 1 month prior to enrollment.
8. Systemic steroid, anti-VEGF or pro-VEGF treatment within 4 months prior to enrollment or anticipated use during the study. These drugs cannot be used during the study.
9. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 9 months. Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed.
10. Individual is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the next 9 months.

The following exclusions apply to the study eye only (i.e., they may be present for the non-study eye unless otherwise specified):

1. Macular edema is considered to be due to a cause other than DME. An eye should not be considered eligible if: (1) the macular edema is considered to be related to ocular surgery such as cataract extraction or (2) clinical exam and/or OCT suggest that vitreoretinal interface abnormalities (e.g., a taut posterior hyaloid or epiretinal membrane) are the primary cause of the macular edema.
2. An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, non-retinal condition, etc.).
3. An ocular condition is present (other than DME) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.).
4. Substantial posterior capsule opacity that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., opacity would be reducing acuity to 20/40 or worse if eye was otherwise normal).
5. History of intravitreal anti-VEGF drug within 21 days prior to enrollment.
6. History of intravitreal or peribulbar corticosteroids within 3 months prior to enrollment.
7. History of macular laser photocoagulation within 4 months prior to enrollment.
8. History of panretinal (scatter) photocoagulation (PRP) within 4 months prior to enrollment or anticipated need for PRP in the 6 months following enrollment into run-in phase.
9. Any history of vitrectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (56):
- United States (56):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Atlantis Eye Care, Huntington Beach, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - California Retina Consultants, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Group of New England, New London, Connecticut
  - New England Retina Associates, Norwich, Connecticut
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - University of Florida College of Med., Department of Ophthalmology, Jacksonville, Florida
  - Central Florida Retina Institute, Lakeland, Florida
  - Ocala Eye Retina Consultants, Ocala, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Retina Associates of Florida, P.A., Tampa, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - Medical Associates Clinic, P.C., Dubuque, Iowa
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, P.A., Shawnee Mission, Kansas
  - Elman Retina Group, P.A., Baltimore, Maryland
  - National Eye Institute/National Institutes of Health, Bethesda, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Retina Vitreous Center, Grand Blanc, Michigan
  - Retina Specialists of Michigan, Grand Rapids, Michigan
  - Retina Center, PA, Minneapolis, Minnesota
  - The Retina Institute, St Louis, Missouri
  - The Institute of Ophthalmology and Visual Science (IOVS), Newark, New Jersey
  - MaculaCare, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - University of Rochester, Rochester, New York
  - Charlotte Eye Ear Nose and Throat Assoc, PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Southwest Retina Specialists, Amarillo, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Baylor Eye Physicians and Surgeons, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Associates of Utah, P.C., Salt Lake City, Utah
  - Virginia Retina Center, Leesburg, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Spokane Eye Clinic, Spokane, Washington
  - University of Wisconsin-Madison, Dept of Ophthalmology/Retina Service, Madison, Wisconsin

REFERENCES:
- [Result] Maturi RK, Glassman AR, Liu D, Beck RW, Bhavsar AR, Bressler NM, Jampol LM, Melia M, Punjabi OS, Salehi-Had H, Sun JK; Diabetic Retinopathy Clinical Research Network. Effect of Adding Dexamethasone to Continued Ranibizumab Treatment in Patients With Persistent Diabetic Macular Edema: A DRCR Network Phase 2 Randomized Clinical Trial. JAMA Ophthalmol. 2018 Jan 1;136(1):29-38. doi: 10.1001/jamaophthalmol.2017.4914. PMID 29127949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 2 multi center randomized trial conducted at 40 US sites; 129 eyes (116 adults) with diabetes between February 2014 and December 2016. Participants with 2 study eyes enrolled one eye in each arm. Therefore, each arm includes no more than 1 study eye per participant; thus the number of eyes is equal to the number of participants in each arm.
Pre-assignment Details: A 12-week run-in phase was conducted to confirm that eyes with persistent diabetic macular edema (DME) still persisted after additional anti-vascular endothelial growth factor (VEGF) injections. At week 12 of the run-in phase, eyes that had received all run-in injections, and continued to meet specific criteria were eligible for randomization.
Units Other Than Participants: Eyes
Groups:
- Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg: The initial intravitreal ranibizumab injection will be given on the day of randomization. The dexamethasone intravitreal injection will be given within 0-8 days of the ranibizumab injection. If defined criteria are met, a second dexamethasone injection in combination with intravitreal ranibizumab (within 0-8 days) will be given at the 12 week visit. If the injections are given consecutively on the same day, the ranibizumab injection must be given first.
  intravitreal ranibizumab 0.3 mg: Intravitreal injection of 0.3mg ranibizumab performed on the day of randomization and up to every 4 weeks using defined treatment criteria. Dexamethasone intravitreal implant: The dexamethasone intravitreal injection will be given within 0-8 days of the ranibizumab injection. If defined criteria are met, a second dexamethasone injection in combination with intravitreal ranibizumab (within 0-8 days) will be given at the 12 week visit. If the injections are given consecutively on the same day, the ran
Period: Overall Study
Arm/Group | Sham + Intravitreal Ranibizumab 0.3 mg | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg
Started (Units in Eyes) | 65; 65 Eyes | 64; 64 Eyes
Completed | 63; 63 Eyes | 64; 64 Eyes
Not Completed | 2; 2 Eyes | 0; 0 Eyes
Not completed — Eyes did not complete or were dropped | 2 | 0

BASELINE CHARACTERISTICS:
Population: Units in Eyes
Units Other Than Participants: Eyes
Groups:
- Sham + Intravitreal Ranibizumab 0.3 mg: Sham and ranibizumab, 0.3 mg, injections
- Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg: Combination of ranibizumab, 0.3 mg and intravitreous sustained dexamethasone drug-delivery system (Ozurdex; Allergan), 700 µg, injection
- Total: Total of all reporting groups
Arm/Group | Sham + Intravitreal Ranibizumab 0.3 mg | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg | Total
Number analyzed (Participants) | 64 | 65 | 116
Number analyzed (Eyes) | 64 | 65 | 129
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 66 [59 to 71] | 64 [59 to 69] | 65 [59 to 70]
Sex/Gender, Customized [Count of Units; unit: Eyes]
  Women | 36 | 31 | 67
  Male | 28 | 34 | 62
Race/Ethnicity, Customized [Count of Units; unit: Eyes]
  White | 35 | 39 | 74
  Black/African American | 9 | 6 | 15
  Hispanic or Latino | 16 | 13 | 29
  Asian | 2 | 6 | 8
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Unknown/not reported | 1 | 1 | 2
Diabetes Type [Count of Units; unit: Eyes]
  Type 1 | 2 | 2 | 4
  Type 2 | 61 | 62 | 123
  Uncertain | 1 | 1 | 2
Duration of Diabetes [Median (Inter-Quartile Range); unit: years] | 19 [10 to 26] | 15 [10 to 21] | 17 [10 to 24]
Insulin Used [Count of Participants; unit: Participants] | 39 | 40 | 79
Hemoglobin A1c [Median (Inter-Quartile Range); unit: Percent Hemoglobin] | 7.4 [6.6 to 8.2] | 7.1 [6.4 to 8.3] | 7.3 [6.5 to 8.2]
Arterial Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 98 [87 to 106] | 97 [87 to 106] | 97 [87 to 106]
Smoking status [Count of Units; unit: Eyes]
  Never | 43 | 44 | 87
  Prior | 14 | 18 | 32
  Current | 7 | 3 | 10
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m˄2] | 33 [29 to 37] | 32 [29 to 37] | 32 [29 to 37]
Participants with 2 study eyes [Number; unit: participants] | 13 | 13 | 26
Prior macular laser treatment for DME [Number; unit: Eyes] | 31 | 31 | 62
Prior Anti-VEGF for DME [Number; unit: Eyes]
  Aflibercept only | 8 | 7 | 15
  Bevacizumab only | 49 | 48 | 97
  Ranibizumab only | 6 | 3 | 9
  Both aflibercept and bevacizumab | 0 | 4 | 4
  Both aflibercept and ranibizumab | 0 | 1 | 1
  Both bevacizumab and ranibizumab | 1 | 2 | 3
Total anti-VEGF injections for DME within the 20 weeks before run-in phase [Median (Inter-Quartile Range); unit: Injections] | 3 [3 to 4] | 3 [3 to 4] | 3 [3 to 4]
Randomization visual acuity letter score [Mean (Standard Deviation); unit: units on a scale] — Best-corrected visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the early treatment diabetic retinopathy study method . Best value on the scale 97, worst 0.
  units on a scale | 63 (13) | 63 (12) | 63 (12)
Randomization central subfield thickness [Mean (Standard Deviation); unit: Microns] — on optical coherence tomography
  Microns | 396 (122) | 375 (97) | 385 (110)
Change in central subfield thickness from enrollment to randomization [Mean (Standard Deviation); unit: Microns] | -50 (102) | -58 (83) | -54 (93)
Improvement in visual acuity(VA) and OCT CST thickness during run-in phase [Number; unit: Eyes] — OCT = Optical coherence tomography CST = Central Subfield Thickness
  Eyes
    Neither VA nor OCT CST is improved | 12 | 15 | 27
    VA and OCT CST are both improved | 22 | 22 | 44
    VA is not improved but OCT CST is improved | 16 | 16 | 32
    VA is improved but OCT CST is not improved | 14 | 12 | 26
Randomization retinal volume [Mean (Standard Deviation); unit: mm3] | 8.6 (2.0) | 8.3 (1.6) | 8.5 (1.8)
Randomization diabetic retinopathy severity level on clinical examination [Number; unit: Eyes] — PDR= Proliferative diabetic retinopathy; NPDR= Non-proliferative diabetic retinopathy
  Eyes
    Mild/moderate NPDR | 28 | 30 | 58
    Severe NPDR | 12 | 10 | 22
    PDR and/or prior scatter laser | 24 | 25 | 49
Change in visual acuity letter score from enrollment to randomization [Mean (Standard Deviation); unit: units on a scale] — Best-corrected visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the early treatment diabetic retinopathy study method. Best value on the scale 97, worst 0.
  units on a scale | 3 (7) | 3 (6) | 3 (7)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity Letter Score
Description: At 24 weeks after randomization, mean change in visual acuity letter score, adjusted for visual acuity at time of randomization
Time Frame: 24 weeks after randomization
Measure: Mean (Standard Deviation); unit: Letter Score
Units Other Than Participants: Eyes
Groups:
- Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg: The initial intravitreal ranibizumab injection will be given on the day of randomization. The dexamethasone intravitreal injection will be given within 0-8 days of the ranibizumab injection. If defined criteria are met, a second dexamethasone injection in combination with intravitreal ranibizumab (within 0-8 days) will be given at the 12 week visit. If the injections are given consecutively on the same day, the ranibizumab injection must be given first. Intravitreal ranibizumab 0.3 mg: Intravitreal injection of 0.3mg ranibizumab performed on the day of randomization and up to every 4 weeks using defined treatment criteria
  dexamethasone intravitreal implant: The dexamethasone intravitreal injection will be given within 0-8 days of the ranibizumab injection. If defined criteria are met, a second dexamethasone injection in combination with intravitreal ranibizumab (within 0-8 days) will be given at the 12 week visit. If the injections are given consecutively on the same day, the ran
Arm/Group | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg | Sham + Intravitreal Ranibizumab 0.3 mg
Number analyzed (Participants) | 63 | 64
Number analyzed (Eyes) | 63 | 64
Letter Score | 2.7 (9.8) | 3.0 (7.1)

2. Secondary Outcome: At 24 Weeks After Randomization, Number of Eyes With at Least 10 and at Least 15 Letter Gain (Increase) or Loss (Decrease) in E-ETDRS Letter Score Visual Acuity.
Description: ETDRS (Early Treatment Diabetic Retinopathy Study)
Time Frame: 24 weeks weeks after randomization
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg | Sham + Intravitreal Ranibizumab 0.3 mg
Number analyzed (Participants) | 63 | 64
Number analyzed (Eyes) | 63 | 64
Eyes
  >= 15 Letter Improvement | 7 | 1
  >= 10 Letter Improvement | 14 | 9
  >= 10 Letter Worsening | 8 | 4
  >= 15 Letter Worsening | 4 | 3

3. Secondary Outcome: Visual Acuity Area Under the Curve (AUC) Between Randomization and 24 Weeks
Description: Only included participants who completed the 24-week visit. Time points for which data were collected for this analysis include 0, 4 8,12, 16, 20, and 24 weeks post randomization.
Time Frame: 24 weeks after randomization
Measure: Mean (Standard Deviation); unit: Letter Score
Units Other Than Participants: Eyes
Arm/Group | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg | Sham + Intravitreal Ranibizumab 0.3 mg
Number analyzed (Participants) | 63 | 64
Number analyzed (Eyes) | 63 | 64
Letter Score | 1.9 (6.3) | 2.5 (4.4)

4. Secondary Outcome: Mean Change in OCT CSF Thickness, Adjusted for Thickness at Time of Randomization
Description: Change in optical coherence tomography (OCT) central subfield thickness (in microns) was truncated to 3 standard deviations from the mean [-372, +201] (calculated using observed changes at 24 weeks combining all treatment groups), to minimize the effect of outliers. Two values were truncated in the sham + ranibizumab group: one on the negative end, and one on the positive end.
Time Frame: 24 weeks after randomization
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg | Sham + Intravitreal Ranibizumab 0.3 mg
Number analyzed (Participants) | 63 | 64
Number analyzed (Eyes) | 63 | 64
microns | -110 (86) | -62 (97)

5. Secondary Outcome: Number of Eyes With ≥1 and ≥2 logOCT Step Gain or Loss in CSF Thickness
Description: Change in optical coherence tomography (OCT) central subfield (CSF) thickness (in microns) was truncated to 3 standard deviations from the mean [-372, +201] (calculated using observed changes at 24 weeks combining all treatment groups), to minimize the effect of outliers. Two values were truncated in the sham + ranibizumab group: one on the negative end, and one on the positive end.
Time Frame: 24 weeks after randomization
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg | Sham + Intravitreal Ranibizumab 0.3 mg
Number analyzed (Participants) | 63 | 64
Number analyzed (Eyes) | 63 | 64
Eyes
  >=1 LogOCT step improvement | 34 | 22
  >= 2 LogOCT step improvement | 14 | 8
  >=1 LogOCT step worsening | 0 | 1
  >=2 LogOCT step worsening | 0 | 1

6. Secondary Outcome: Eyes With OCT CSF Thickness < the Gender-specific Spectral Domain OCT Equivalent of 250 Microns on Zeiss Stratus
Description: Gender and OCT machine-specific values for OCT central subfield thickness (in microns) are defined as: <290 in women and <305 in men in Zeiss Cirrus; <305 in women and <320 in men in Heidelberg Spectralis
Time Frame: 24 weeks after randomization
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg | Sham + Intravitreal Ranibizumab 0.3 mg
Number analyzed (Participants) | 63 | 64
Number analyzed (Eyes) | 63 | 64
Eyes | 32 | 20

7. Secondary Outcome: OCT CSF Thickness Area Under the Curve Between Randomization and 24 Weeks
Description: Including participants who completed the 24-week visit. Time points for which data were collected for this analysis include 0, 4 8,12, 16, 20, and 24 weeks post randomization.
Time Frame: 24 weeks after randomization
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg | Sham + Intravitreal Ranibizumab 0.3 mg
Number analyzed (Participants) | 63 | 64
Number analyzed (Eyes) | 63 | 64
microns | -86.9 (65.6) | -33.5 (56.8)

ADVERSE EVENTS:
Time Frame: From Randomization to 24-weeks
Groups:
- Bilateral: Participants with one eye enrolled in each arm of the study. A participant could only have one eye in each arm/group, therefore participants in the bilateral group received Intravitreal dexamethasone+intravitreal ranibizumab 0.3mg in one eye and Sham + intravitreal ranibizumab 0.3 mg in the other eye.
Arm/Group | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg | Sham + Intravitreal Ranibizumab 0.3 mg | Bilateral
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51 | 0/13
Serious Adverse Events (participants affected / at risk) | 7/52 | 7/51 | 1/13
Other Adverse Events (participants affected / at risk) | 38/52 | 29/52 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg (N=52) | Sham + Intravitreal Ranibizumab 0.3 mg (N=51) | Bilateral (N=13)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stent placement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Vascular graft (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Intravitreal Dexamethasone+Intravitreal Ranibizumab 0.3mg (N=52) | Sham + Intravitreal Ranibizumab 0.3 mg (N=52) | Bilateral (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0/51 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1/51 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0/51 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1/51 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1/51 (1) | 0 (0)
Diabetes mellitus inadequate control (Endocrine disorders) | 1 (1) | 0/51 (0) | 0 (0)
Hypoglycaemia (Endocrine disorders) | 0 (0) | 0/51 (0) | 1 (1)
Asthenopia (Eye disorders) | 1 (3) | 0/51 (0) | 0 (0)
Blepharitis (Eye disorders) | 2 (3) | 0/51 (0) | 0 (0)
Cataract (Eye disorders) | 3 (3) | 1/51 (1) | 0 (0)
Cataract cortical (Eye disorders) | 0 (0) | 0/51 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (1) | 0/51 (0) | 2 (2)
Cataract subcapsular (Eye disorders) | 1 (1) | 0/51 (0) | 2 (3)
Conjunctival haemorrhage (Eye disorders) | 4 (4) | 0/51 (0) | 1 (1)
Corneal defect (Eye disorders) | 0 (0) | 0/51 (0) | 1 (1)
Corneal oedema (Eye disorders) | 1 (1) | 0/51 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0/51 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0/51 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1/51 (1) | 1 (2)
Ectropion (Eye disorders) | 1 (1) | 0/51 (0) | 0 (0)
Eye irritation (Eye disorders) | 2 (2) | 1/51 (1) | 0 (0)
Eye pain (Eye disorders) | 2 (2) | 3/51 (3) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 1/51 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1/51 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0/51 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 1/51 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0/51 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0/51 (0) | 1 (1)
Metamorphopsia (Eye disorders) | 0 (0) | 1/51 (1) | 0 (0)
Ocular discomfort (Eye disorders) | 1 (1) | 1/51 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1/51 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1/51 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1/51 (1) | 0 (0)
Retinal exudates (Eye disorders) | 1 (1) | 0/51 (0) | 0 (0)
Vision blurred (Eye disorders) | 7 (7) | 4/51 (5) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 2/51 (3) | 0 (0)
Visual field defect (Eye disorders) | 1 (1) | 0/51 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1/51 (2) | 0 (0)
Vitreous adhesions (Eye disorders) | 0 (0) | 0/51 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 8 (8) | 3/51 (3) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0/51 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1/51 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1/51 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0/51 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0/51 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0/51 (0) | 0 (0)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1) | 0/51 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1/51 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0/51 (0) | 0 (0)
Tooth infection (Gastrointestinal disorders) | 0 (0) | 1/51 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0/51 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2/51 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1/51 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1/51 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2/51 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0/51 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1/51 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0/51 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1/51 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1/51 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1/51 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0/51 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1/51 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0/51 (0) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 1/51 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0/51 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 11 (12) | 0/51 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1/51 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0/51 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1/51 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1/51 (1) | 0 (0)
Foot fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/51 (0) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 0/51 (0) | 1 (1)
Multiple fractures (Musculoskeletal and connective tissue disorders) | 0 (0) | 1/51 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/51 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1/51 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/51 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/51 (0) | 0 (0)
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0/51 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1/51 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0/51 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1/51 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0/51 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1/51 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0/51 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0/51 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1/51 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1/51 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0/51 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1/51 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0/51 (0) | 2 (2)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2/51 (2) | 1 (1)
Pharyngitis streptococcal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0/51 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1/51 (2) | 0 (0)
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0/51 (0) | 1 (1)
Skin cancer (Skin and subcutaneous tissue disorders) | 0 (0) | 0/51 (0) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0/51 (0) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 1/51 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 2 (3) | 0/51 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0/51 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial results can not be discussed until they have been made available to the public

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT01945866/SAP_000.pdf
  • Study Protocol (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT01945866/Prot_001.pdf